CLINICAL TRIAL: NCT04918082
Title: Assessment of Quality of Life and Treatment Times for Patients With Invasive Type Breast Cancer in Martinique
Acronym: Qualibreast-MQ
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Other Study IDs: 20_RIPH3_06; 2020-A01290-39 (Other: DGS, Ministry of Health)
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Breast Neoplasms; Quality of Life; Survivorship
Keywords: Breast cancer; Quality of life; Survivorship; Survival; French West Indies
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Quality of life questionnaires — Patients' quality of life will be assessed with self-reported items through both the EORTC-QLQ-C30 and EORTC-QLQ-BR23 modules.

SUMMARY:
Cancer and its treatments can be factors that alter the quality of life of patients. The induced alteration of the quality of life can influence compliance and impact survival. Considering the after-effects of the treatment, carrying out such a survey will provide for the first time precise information on the main determinants of the quality of life as well as on the care pathway of patients with invasive breast cancer in the Martinique region.

DETAILED DESCRIPTION:
Breast cancer is the second most common cancer in the West Indies and the leading cancer in women. With 215 new cases in Guadeloupe, 204 in Martinique and 56 in French Guiana each year, it accounts for 37%, 33% and 26% of incident cancer cases in women respectively, but also affects men. Its incidence, lower than in France, is increasing over the period 2008-2014. The diagnostic and therapeutic management of cancer can have an impact on the quality of life of patients, taking into account the adverse effects occurring during and after treatment, both in the short and long term. The European Organisation for Research and Treatment of Cancer (EORTC) has developed a series of questionnaires to assess the quality of life of cancer patients, including a general questionnaire (QLQ-C30) and specific modules for breast cancer (EORTC BREAST (EORTC QLQ-BR23)) with the objective of improving professional practices.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age residing in Martinique with invasive breast cancer diagnosed from 2020 (single tumor at diagnosis)
* Patients who have read the information note and have indicated that they do not wish to participate in the study
* Patient with social security coverage.

Exclusion Criteria:

* Refusal to participate
* Patient with insitu breast cancer
* Patient with a second cancer
* Patient with cancer within 5 years prior to inclusion
* Patient who could not answer quality of life questionnaires
* Patient not fluent in French
* Person under legal protection (safeguard of justice, guardianship, curators , etc.).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breast cancer followed at the Martinique University Hospital
Sampling Method: Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2025-12-28 (Estimated); Study Completion 2026-06-28 (Estimated)

PRIMARY OUTCOMES:
Assessment of global disorders in patients with breast cancer | 12 months after diagnosis
  Quality of life of patients with invasive breast cancer in Martinique assessed by QLQ-C30
Assessment of disorders specific to breast cancer patients Assessment of disorders specific to breast cancer patients | 12 months after diagnosis
  Quality of life of patients with invasive breast cancer in Martinique assessed by QLQ-BR23
Assessment of global disorders in patients with breast cancer | 36 months after diagnosis
  Quality of life of patients with invasive breast cancer in Martinique assessed by QLQ-C30
Assessment of disorders specific to breast cancer patients | 36 months after diagnosis
  Quality of life of patients with invasive breast cancer in Martinique assessed by QLQ-BR23

CONTACTS AND LOCATIONS:
Overall Officials: Clarisse JOACHIM-CONTARET, Principal Investigator — CHU Martinique
Locations (1):
- CHU Martinique, Fort-de-France, Martinique